CLINICAL TRIAL: NCT00914979
Title: AngioSculpt Scoring Balloon Catheter For Bifurcation Coronary Lesions (ABC Study) Prospective, Multi-center, Non-randomized, Single-arm Registry
Brief Title: AngioSculpt Scoring Balloon Catheter For Bifurcation Coronary Lesions (ABC Study)
Acronym: ABC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties in recruiting patients
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0033 - 08 - EMC
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Bifurcation Coronary Disease
Keywords: Angiosculpt; Bifurcation Lesion; Side branch; IVUS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Single Arm - Interventional
  Interventions: Device: AngioSculpt

INTERVENTIONS:
Device: AngioSculpt — The AngioSculpt Scoring Balloon Catheter is a standard balloon dilatation catheter with a scoring balloon near the distal tip

SUMMARY:
Assess the impact of lesion preparation using the AngioSculpt balloon in the treatment of bifurcation lesions in native coronary arteries.

DETAILED DESCRIPTION:
The purpose of the AngioSculpt® Scoring Balloon Catheter For Bifurcation Coronary lesions (ABC registry) is to demonstrate the acute procedural success, device performance and long term outcome associated with use of the AngioSculpt Scoring Balloon Catheter (AngioScore, Inc., Fremont, CA) for lesion preparation in the treatment of bifurcation lesions in native coronary arteries

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant (≥ 50% diameter stenosis) native coronary artery disease involving a bifurcation (Medina class (x,x,1)).

Exclusion Criteria:

* Concomitant use of Rotablator, Cutting Balloon, or investigational coronary devices.
* Additional planned coronary interventions for a non-target lesion within 30 days of the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Procedural success ≤ 50% diameter stenosis of the main and the side branch at the conclusion of the procedure in the absence of in-hospital MACE | 9 Months

SECONDARY OUTCOMES:
Rate of side branch stenting | 9 Months
Angiographic dissection rate and grade | 9 months
MACE rate at 30 days post-procedure | 9 months
Cumulative stent thrombosis and TLR rates at 9 months | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Suleiman, MD, Principal Investigator — Heart Institute; Ha'Emek Medical Center
Locations (4):
- Israel (4):
  - Khalid Suleiman, Afula
  - Oded Izenberg, Rehovot
  - Alexander Goldberg, Safed
  - Ricardo Krakover, Zrifin